CLINICAL TRIAL: NCT05743712
Title: A Mobile Text Approach to Measurement and Feedback for Wraparound Care Coordination
Brief Title: Pilot Test of a Mobile Text Approach to Measurement and Feedback for Wraparound Care Coordination
Acronym: SMART-Wrap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3CG079Pilot
Record Dates: First submitted 2023-02-07; First posted 2023-02-24 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Mental Health Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART-Wrap (Experimental): SMART-Wrap is a prototype measurement and feedback software system tailored to Wraparound service model (WSM) for emotional disorders to provide measurement-based care in care coordination for youth behavioral health.
  Interventions: Other: SMART-Wrap

INTERVENTIONS:
Other: SMART-Wrap — This intervention, SMS (short message system)-based augmentation, seeks to improve the impact and approach of the Wraparound service model by utilizing SMS, which has been shown to increase treatment adherence and sustained engagement. This intervention will facilitate regular, repeated evaluation of intermediate outcomes through self-report assessments.

SUMMARY:
This SBIR Phase I study will test the acceptability and feasibility of a novel measurement and feedback system tailored to Wraparound service model (WSM) for emotional disorders to produce a feasible, cost-efficient, and scalable software system to meet the pressing public health need for Measurement-based Care in care coordination for youth behavioral health.

DETAILED DESCRIPTION:
The goal of this SBIR is to test a novel mobile and text-based measurement and feedback system tailored to WSM. Investigators will recruit 10 care teams (50 care team members total: 10 managers/administrators, 10 supervisors, and 30 care coordinators), 30 caregivers, and 15 youth/young adults (14+ yo) with SED currently enrolled in WSM. Caregivers of minor children aged 5-17 and caregivers of young adults 18-26 will be invited to participate. However, only parents with youth aged 14-17 will be invited to consider participation for their children, as well, and young adults age 18-26 will have the opportunity to participate without a caregiver If a caregiver has multiple children enrolled in Wraparound, we will select one child to invite to participate. Of those eligible, investigators will select 30 caregivers and up to 15 youth/young adults (14+) that have access to a mobile device. These participants will be informed of the project by members of their care team and asked to complete a consent to contact if they are interested in learning more about the research study. Interested families will be asked to review consent materials and sign up online. Caregivers and youth/young adults will participate in a 30-minute study orientation meeting and then interact independently with the system over a 4-week period. During this time, care team members will have access to the SMART-Wrap website, where they can view the survey feedback from their families. Care team members will be expected to interact with the system throughout the test period and may adjust care based on the feedback they receive. Within 5 days of the last text message, caregivers and youth/young adults will complete a brief survey evaluating the prototype in the following areas of usability, acceptability, and feasibility, as well as complete the 10-item System Usability Survey (SUS). Care team members will complete a similar survey that asks about these same areas, but also includes items about compatibility with existing wraparound treatment planning and implementation, interoperability with existing electronic record management systems, duplicative vs. complementary with existing systems, and added value over existing methods. Following completion of their evaluation, participants will be invited to take part in 45-minute interviews or virtual focus groups (separately for care team members, caregivers, and youth/young adults). Of the participants that agree, 10 care team members, 10 caregivers, and 10 youth/young adults will be selected to complete the virtual focus group.

ELIGIBILITY:
Inclusion Criteria:

* Wraparound Service Model Care teams (each consisting of 1 manager or administrator, 1 supervisor, and up to 3 care coordinators) must coordinate the care of one youth/young adult (ages 5-26).
* Wraparound Service Model enrolled families can consist of either (a) a caregiver of a youth/young adult age 5-26 (participating without their child), (b) a caregiver of a youth/young adult age 14-26 (participating with their child - adult children sign separate consent to contact forms and enroll separately), or (c) a young adult age 18-26 participating without their caregiver.

Exclusion Criteria:

* youth/young adults known to providers to have expressed risk of harm to themselves or others within the 6 months prior to the recruitment period

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Prototype Evaluation for Families | 5-week follow-up post messaging protocol
  Caregivers, youth, and young adults will complete this 12-item measure, rating the extent to which they agree with statements about the usability, acceptability, and feasibility of the SMART-Wrap system. The measure includes 9 Likert items and 3 open-ended items. Responses to the Likert items range from 1 (Completely Disagree) to 5 (Completely Agree). Total scores are based on the Likert items are range from 0 to 45. Higher scores reflect more positive opinions.
Prototype Evaluation for Care Team Members | 5-week follow-up post messaging protocol
  Care team members will complete this 34-item measure, rating the extent to which they agree with statements about the SMART-Wrap system. The measure includes 7 open-ended items, one yes/no item, and 26 Likert-scale items about the usability, acceptability, and feasibility of the system, and items about the system's interoperability with existing electronic record management systems, whether it is duplicative or complementary with existing systems, and its added value over existing methods of collecting feedback from families in Wraparound. Responses to the Likert items range from 1 (Completely Disagree) to 5 (Completely Agree). Total scores are based on the Likert items and range from 0 to 130. Higher scores reflect more positive opinions.
System Usability Survey | 5-week follow-up post messaging protocol
  Caregivers, youth, young adults, and care team members will complete this 10-item measure, rating the extent to which they agree with statements about the usability of the SMART-Wrap system. Responses range from 1 (Completely Disagree) to 5 (Completely Agree). For items 1, 3, 5, 7, and 9, higher scores reflect more positive outcomes. For items 2, 4, 6, 8, and 10, higher scores reflect more negative outcomes. Items 2, 4, 6, 8, and 10 are reverse coded, and all survey items are rescaled from 0 to 4 and multiplied by 2.5 to calculate total scores, which range from 0 to 100.

SECONDARY OUTCOMES:
Results from Caregiver Text Message Items | 4-item sets of survey items administered weekly over a 4-week period
  Caregivers will complete this 16-item measure, rating the extent to which they agree with statements about therapeutic alliance with their Wraparound care team, their satisfaction with Wraparound, the care team's fidelity to the Wraparound care model, and their outcomes because of participating in Wraparound. Responses range from 0 (Not at All) to 4 (Absolutely). Total scores range from 0 to 64. Higher scores reflect greater satisfaction, therapeutic alliance, and fidelity and better outcomes.
Results from Youth Text Message Items | 2-item sets of surveys items administered weekly over a 4-week period
  Youth and young adults will complete this 8-item measure, rating the extent to which they agree with statements about their satisfaction with Wraparound and their outcomes as a result of participating in Wraparound. Responses range from 0 (Not at All) to 4 (Absolutely). Total scores range from 0 to 32. Higher scores reflect greater satisfaction and better outcomes.
Usage Metrics from the SMART-Wrap system for families | 4-week period
  The SMART-Wrap software will track whether each text message is opened, the length of time between delivery and opening, and length of time between opening and submission of item response. These metrics are measured in seconds. In all cases, a shorter time span indicates more positive outcomes.
Usage Metrics from the SMART-Wrap system for care team members | the period in which any families served by the care team are interacting with the SMART-Wrap system, approximately 8-weeks
  The SMART-Wrap software will track usage of the SMART-Wrap dashboard by the care team, including number of logins, amount of time spent (in seconds), and number/type of technical assistance requests. Number of logins and number of technical requests are measured as counts. Higher numbers of logins indicates a more positive outcome, higher time spent indicates a more positive outcome, and lower number of technical requests represents a more positive outcome.
Results from focus groups / interviews with families | 45-minutes, completed after the test of the SMART-Wrap system
  10 caregivers and 10 youth/young adults will participate in either focus groups or individual interviews. They will be asked about their experience with the SMART-Wrap system, strengths and weaknesses of SMART-Wrap, and challenges to using SMART-Wrap. Comments will be combined and grouped based on themes in a qualitative summary.
Results from focus groups / interviews with care team members | 45-minutes, completed after the test of the SMART-Wrap system
  10 care team members will participate in either focus groups or individual interviews. They will be asked about strengths and weaknesses of SMART-Wrap, and challenges to using SMART-Wrap, and recommendations for revisions to SMART-Wrap. Comments will be combined and grouped based on themes in a qualitative summary.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa DeRosier, PhD, Principal Investigator — 3C Institute; Eric Bruns, PhD, Principal Investigator — University of Washington
Locations (1):
- 3C Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No